CLINICAL TRIAL: NCT00751348
Title: Immunogenicity & Safety Study of GSK Biologicals' Combined Measles-mumps-rubella-varicella Vaccine 208136
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 110876
Record Dates: First submitted 2008-09-10; First posted 2008-09-11 (Estimated); Results first posted 2017-04-24 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2017-05

CONDITIONS: Measles; Varicella; Mumps; Rubella
Keywords: second year of life; one-dose schedule; varicella; rubella; measles; mumps
MeSH Terms: conditions — Measles; Chickenpox; Mumps; Rubella | interventions — Priorix-Tetra vaccine

ARMS (2):
- PRIORIX-TETRA GROUP (Experimental): Healthy male and female subjects between, and including 11 and 24 months of age, who received one dose of Priorix-Tetra® vaccine at Day 0, administered subcutaneously in the deltoid region of the left upper arm.
  Interventions: Biological: Priorix-Tetra®
- PRIORIX + VARILRIX GROUP (Active Comparator): Healthy male and female subjects between, and including 11 and 24 months of age, who received one dose of Priorix™ vaccine together with one dose of Varilrix™ vaccine at Day 0, administered subcutaneously in the deltoid regions of the left or right upper arm, respectively.
  Interventions: Biological: PriorixTM; Biological: VarilrixTM

INTERVENTIONS:
Biological: PriorixTM — Subcutaneous administration in left upper arm
  Arms: PRIORIX + VARILRIX GROUP
Biological: VarilrixTM — Subcutaneous administration in right upper arm
  Arms: PRIORIX + VARILRIX GROUP
Biological: Priorix-Tetra® — Subcutaneous injection in left upper arm
  Arms: PRIORIX-TETRA GROUP

SUMMARY:
This Phase 3b study is being conducted for the purpose of registration of the GSK208136 vaccine in Korea.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female between, and including 11 and 24 months of age, at the time of the vaccination.
* Written informed consent obtained from the parent or guardian of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the vaccine dose.
* Administration of immunoglobulins and/or any blood products during the six months before entering the study or planned administration during the study period.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within 30 days prior to until 42 days after the study vaccine dose with the exception of inactivated vaccines such as pneumococcal, Haemophilus influenzae type b conjugate vaccines, inactivated influenza, hepatitis A or B vaccine or diphtheria/tetanus-containing vaccines which can be administered up to eight days before the study vaccine dose.
* Previous vaccination against measles, mumps, rubella and/or varicella.
* History of measles, mumps, rubella and/or varicella/zoster diseases.
* Known exposure to measles, mumps, rubella and/or varicella within 30 days prior to study start.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* A family history of congenital or hereditary immunodeficiency.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine(s), including systemic hypersensitivity to neomycin.
* Major congenital defects or serious chronic illness.
* Acute disease at the time of enrolment.
* Rectal temperature ≥ 38°C or axillary temperature ≥ 37.5°C at the time of vaccination.
* Residence in the same household as a high risk person e.g.:
* New-born infants (0-4 weeks of age)
* Pregnant women who have a negative history of chickenpox
* Persons with known immunodeficiency

Ages: 11 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 475 (Actual)
Dates: Start 2008-10-01; Primary Completion 2010-05-27 (Actual); Study Completion 2010-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (11):
- South Korea (11):
  - GSK Investigational Site, Bucheon-si
  - GSK Investigational Site, Daejeon
  - GSK Investigational Site, Gwangju
  - GSK Investigational Site, GyeongSangNam-do
  - GSK Investigational Site, Iksan
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Jeonju Jeonbuk
  - GSK Investigational Site, Seongnam-si, Gyeonggi-do
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Uijeongbu, Kyonggi-do
  - GSK Investigational Site, Wonju-si Kangwon-do

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Cha SH, Shin SH, Lee TJ, Kim CH, Povey M, Kim HM, Nicholson O. Immunogenicity and safety of a tetravalent measles-mumps-rubella-varicella vaccine: an open-labeled, randomized trial in healthy Korean children. Clin Exp Vaccine Res. 2014 Jan;3(1):91-9. doi: 10.7774/cevr.2014.3.1.91. Epub 2013 Dec 18. PMID 24427766
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 110876 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110876 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 110876 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 110876 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 110876 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 110876 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of 475 subjects enrolled in the study, one did not receive any vaccination.
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Period: Overall Study
Arm/Group | Priorix-Tetra Group | Priorix + Varilrix Group
Started | 313 | 161
Completed | 307 | 159
Not Completed | 6 | 2
Not completed — Withdrawal by Subject | 5 | 2
Not completed — Migration from study area | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Priorix-Tetra Group | Priorix + Varilrix Group | Total
Number analyzed (Participants) | 313 | 161 | 474
Age, Continuous [Mean (Standard Deviation); unit: Months] | 12.4 (1.4) | 12.5 (1.65) | 12.43 (1.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 76 | 204
  Male | 185 | 85 | 270
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian-East Asian Heritage | 313 | 159 | 472
  Asian-South East Asian Heritage | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Seroconverted for Measles, Mumps, Rubella and Varicella Zoster Virus (VZV) Antibodies Above the Cut-off Values
Description: Seroconversion was defined as the appearance of antibodies [i.e. titer greater than or equal to (≥) the cut-off value] in the sera of subjects seronegative [i.e. titer below (<) cut-off value] before vaccination. Cut-off values were the following: Anti-measles concentration ≥ 150 milli-international units per milliliter (mIU/mL); Anti-mumps concentration ≥ 231 units per milliliter (U/mL); Anti-rubella concentration ≥ 4 international units per milliliter (IU/mL); Anti-VZV titer ≥ 1:4 dilution.
Time Frame: At 42 days post-vaccination
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity,which included all evaluable subjects who were seronegative for at least one vaccine antigen at baseline and for whom pre-vaccination and post-vaccination serology results were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Priorix-Tetra Group | Priorix + Varilrix Group
Number analyzed (Participants) | 300 | 157
Participants
  Anti-Measles: number analyzed (Participants) | 300 | 156
  Anti-Measles | 294 | 155
  Anti-Mumps: number analyzed (Participants) | 295 | 154
  Anti-Mumps | 262 | 145
  Anti-Rubella: number analyzed (Participants) | 298 | 157
  Anti-Rubella | 297 | 157
  Anti-VZV: number analyzed (Participants) | 283 | 151
  Anti-VZV | 280 | 151
Statistical Analysis 1: Comparison: Priorix-Tetra Group vs Priorix + Varilrix Group; Non-inferiority of Priorix-Tetra® vaccine vs Priorix™ and Varilrix™ administered as concomitant vaccine 42-56 days after vaccination at Day 0 in terms of anti-measles seroconversion rates; Test type: Non-Inferiority — Criterion for evaluation of non-inferiority: the lower limit (LL) of the two-sided standardized asymptotic 95% confidence interval (CI) for the group difference (Priorix-Tetra Group minus Priorix+Varilrix Group) in seroconversion rate for anti-measles was above -10%; p < 0.05, Fisher Exact — The P-value for all reactogenicity comparisons was below (<) 0.05; Difference in percentage = -1.36, 95% CI 2-sided [-3.77 to 1.66]
Statistical Analysis 2: Comparison: Priorix-Tetra Group vs Priorix + Varilrix Group; Non-inferiority of Priorix-Tetra® vaccine vs Priorix™ and Varilrix™ administered as concomitant vaccine 42-56 days after vaccination at Day 0 in terms of anti-mumps seroconversion rates; Test type: Non-Inferiority — Criterion for evaluation of non-inferiority: the lower limit (LL) of the two-sided standardized asymptotic 95% confidence interval (CI) for the group difference (Priorix-Tetra Group minus Priorix+Varilrix Group) in seroconversion rate for anti-mumps was above -10%; p < 0.05, Fisher Exact — The P-value for all reactogenicity comparisons was below (<) 0.05; Difference in percentage = -5.34, 95% CI 2-sided [-10.4 to 0.38]
Statistical Analysis 3: Comparison: Priorix-Tetra Group vs Priorix + Varilrix Group; Non-inferiority of Priorix-Tetra® vaccine vs Priorix™ and Varilrix™ administered as concomitant vaccine 42-56 days after vaccination at Day 0 in terms of anti-rubella seroconversion rates; Test type: Non-Inferiority — Criterion for evaluation of non-inferiority: the lower limit (LL) of the two-sided standardized asymptotic 95% confidence interval (CI) for the group difference (Priorix-Tetra Group minus Priorix+Varilrix Group) in seroconversion rate for anti-rubella was above -10%; p < 0.05, Fisher Exact — The P-value for all reactogenicity comparisons was below (<) 0.05; Difference in percentage = -0.34, 95% CI 2-sided [-1.88 to 2.06]
Statistical Analysis 4: Comparison: Priorix-Tetra Group vs Priorix + Varilrix Group; Non-inferiority of Priorix-Tetra® vaccine vs Priorix™ and Varilrix™ administered as concomitant vaccine 42-56 days after vaccination at Day 0 in terms of anti-varicella zoster virus (anti-VZV) seroconversion rates; Test type: Non-Inferiority — Criterion for evaluation of non-inferiority: the lower limit (LL) of the two-sided standardized asymptotic 95% confidence interval (CI) for the group difference (Priorix-Tetra Group minus Priorix+Varilrix Group) in seroconversion rate for anti-VZV was above -10%; p < 0.05, Fisher Exact — The P-value for all reactogenicity comparisons was below (<) 0.05; Difference in percentage = -1.06, 95% CI 2-sided [-3.07 to 1.44]

2. Secondary Outcome: Antibody Concentrations Against Measles
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs), expressed in milli-international units per milliliter (mIU/mL).
Time Frame: At 42-days post-vaccination
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects who were seronegative for at least one vaccine antigen at baseline and for whom pre-vaccination and post-vaccination serology results were available.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Priorix-Tetra Group | Priorix + Varilrix Group
Number analyzed (Participants) | 300 | 156
mIU/mL | 4978.6 [4579.8 to 5412.1] | 3433.6 [3116.3 to 3783.2]

3. Secondary Outcome: Antibody Concentrations Against Mumps
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs), expressed in units per milliliter (U/mL).
Time Frame: At 42-days post-vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | Priorix-Tetra Group | Priorix + Varilrix Group
Number analyzed (Participants) | 295 | 154
U/mL | 1012.3 [894.4 to 1145.7] | 934.3 [805.2 to 1084.1]

4. Secondary Outcome: Antibody Concentrations Against Rubella
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs), expressed in international units per milliliter (IU/mL).
Time Frame: At 42-days post-vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Priorix-Tetra Group | Priorix + Varilrix Group
Number analyzed (Participants) | 298 | 157
IU/mL | 63.4 [57.9 to 69.4] | 75.7 [68 to 84.3]

5. Secondary Outcome: Antibody Titers Against Varicela Viruses
Description: Antibody titers were presented as geometric mean titers (GMTs).
Time Frame: At 42-days post-vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Priorix-Tetra Group | Priorix + Varilrix Group
Number analyzed (Participants) | 283 | 151
Titers | 134.1 [117 to 153.7] | 129.2 [109.8 to 152]

6. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Solicited local symptoms assessed were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = cry when limb was moved/spontaneously painful. Grade 3 redness/swelling = redness/swelling spreading beyond 20 millimeters (mm) of injection site.
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects who had their symptoms sheet filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | Priorix-Tetra Group | Priorix + Varilrix Group
Number analyzed (Participants) | 310 | 159
Participants
  Any Pain | 15 | 10
  Grade 3 Pain | 0 | 0
  Any Redness | 26 | 21
  Grade 3 Redness | 0 | 1
  Any Swelling | 5 | 5
  Grade 3 Swelling | 0 | 0

7. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Solicited general symptoms assessed were fever [defined as rectal temperature ≥38.0 degrees Celsius (°C)], rash, meningism and parotid gland swelling. Any= incidence of the specified symptoms regardless of intensity grade or relationship to study vaccine. Grade 3 fever= rectal temperature above (>) 39.5°C. Grade 3 rash= more than 150 lesions. Grade 3 meningism and parotid gland swelling= meningism/parotid gland swelling symptom which prevented normal everyday activities. Related = general symptom assessed by the investigator as causally related to the vaccination.
Time Frame: During the 43-day (Days 0-42) post-vaccination period
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects who had the symptoms sheet filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | Priorix-Tetra Group | Priorix + Varilrix Group
Number analyzed (Participants) | 310 | 159
Participants
  Any Temperature | 202 | 82
  Grade 3 Temperature | 53 | 19
  Related Temperature | 31 | 12
  Any Rash | 33 | 16
  Grade 3 Rash | 0 | 0
  Related Rash | 3 | 1
  Any Meningism | 2 | 0
  Grade 3 Meningism | 0 | 0
  Related Meningism | 0 | 0
  Any Parotid gland swelling | 0 | 0
  Grade 3 Parotid gland swelling | 0 | 0
  Related Parotid gland swelling | 0 | 0

8. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any was defined as an adverse event (AE) reported in addition to those solicited during the clinical study. Any solicited symptom with onset outside the specified period of follow-up for solicited symptoms was reported as an unsolicited adverse event.
Time Frame: Within the 43-day (Days 0-42) post-vaccination period
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Priorix-Tetra Group | Priorix + Varilrix Group
Number analyzed (Participants) | 313 | 161
Participants | 194 | 88

9. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that resulted in death, were life threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: During the entire study period (from Day 0 up to Day 43 or Day 57)
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Priorix-Tetra Group | Priorix + Varilrix Group
Number analyzed (Participants) | 313 | 161
Participants | 25 | 12

ADVERSE EVENTS:
Time Frame: Solicited local: during the 4-day (Days 0-3) post-vaccination period. Solicited general symptoms and unsolicited AEs: during the 43-day (Days 0-42) post-vaccination period. SAEs: during the entire study period (from Day 0 up to Day 43 or 57).
Description: The solicited local and general symptoms were only collected from those subjects who filled in their symptom sheets.
Arm/Group | Priorix-Tetra Group | Priorix + Varilrix Group
All-Cause Mortality (participants affected / at risk) | 0/313 | 0/161
Serious Adverse Events (participants affected / at risk) | 25/313 | 12/161
Other Adverse Events (participants affected / at risk) | 243/313 | 113/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Priorix-Tetra Group (N=313) | Priorix + Varilrix Group (N=161)
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Febrile convulsion (Nervous system disorders) | 2 | 0
Pyrexia (General disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1
Hypophagia (Metabolism and nutrition disorders) | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1
Acute tonsillitis (Infections and infestations) | 1 | 0
Bronchiolitis (Infections and infestations) | 3 | 2
Bronchopneumonia (Infections and infestations) | 6 | 3
Croup infectious (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 5 | 6
Gastroenteritis norovirus (Infections and infestations) | 1 | 0
Gastroenteritis rotavirus (Infections and infestations) | 2 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 1
Herpangina (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Otitis media acute (Infections and infestations) | 3 | 1
Pharyngitis (Infections and infestations) | 5 | 1
Pharyngotonsillitis (Infections and infestations) | 4 | 1
Pneumonia (Infections and infestations) | 1 | 1
Rhinitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Viral rash (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Priorix-Tetra Group (N=313) | Priorix + Varilrix Group (N=161)
Pain (General disorders) | 15/310 | 10/159
Redness (General disorders) | 26/310 | 21/159
Fever (General disorders) | 202/310 | 82/159
Rash (General disorders) | 33/310 | 16/159
Upper respiratory tract infection (Infections and infestations) | 63 | 25
Nasopharyngitis (Infections and infestations) | 31 | 14
Gastroenteritis (Infections and infestations) | 28 | 13
Pharyngitis (Infections and infestations) | 27 | 10
Bronchitis (Infections and infestations) | 26 | 11
Pharyngotonsillitis (Infections and infestations) | 21 | 10
Otitis media acute (Infections and infestations) | 13 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.